CLINICAL TRIAL: NCT07210021
Title: Diagnostic Accuracy, Usability, Patient Compliance, and System Reliability of the AK+ Guard™ ECG Application for Hyperkalemia Prediction in Ambulatory Chronic Kidney Disease Patients (Outpatient and Remote Monitoring Arms)
Brief Title: AK+ Guard™ Pilot Study in Chronic Kidney Disease: Outpatient Diagnostic Accuracy and Remote Monitoring
Status: Recruiting | Type: Observational
Sponsor: AccurKardia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AKG CKD 002A, AKG CKD 002B
Record Dates: First submitted 2025-09-15; First posted 2025-10-07 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hyperkalemia; Chronic Kidney Disease (Stage 3-4)
Keywords: hyperkalemia; ambulatory CKD; CKD; chronic kidney disease; ECG
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For this study, no biospecimens are being collected by the investigators. Rather, the study is collecting ECGs at the time of routine clinical blood draws for serum potassium labs. The study is only retaining the laboratory result for serum potassium. The laboratory is obtaining the serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 2A - Outpatient Diagnostic Accuracy: Participants with chronic kidney disease (CKD) stages III-IV who are scheduled for a routine outpatient potassium blood test. At the same clinic visit, participants will have ECGs recorded using three devices (12-lead ECG, Apple Watch, and HeartBeam) for analysis by the AK+ Guard™ software. Researchers will compare the software's results with the laboratory potassium values to estimate sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).
  Interventions: Device: AK+ Guard™ ECG Application
- Arm 2B - Remote Patient Monitoring: A subset of participants from Arm 2A (Outpatient Diagnostic Accuracy) who agree to continue with at-home monitoring for up to four weeks. These participants will use an Apple Watch and study application to record daily ECGs. They will complete short weekly surveys about ease of use, anxiety, and safety perceptions, and return for a confirmatory laboratory test if the AK+ Guard™ software signals possible high potassium. Researchers will assess daily compliance, usability, and overall system reliability in a real-world setting.
  Interventions: Device: AK+ Guard™ ECG Application

INTERVENTIONS:
Device: AK+ Guard™ ECG Application — An investigational Software as a Medical Device (SaMD) that analyzes Lead I electrocardiogram (ECG) data using artificial intelligence to detect moderate to severe hyperkalemia (serum potassium ≥ 6.5 mmol/L). ECG inputs may be obtained from standard 12-lead ECGs, clinical-grade ECG devices with Lead I capability, or consumer wearable devices (e.g., Apple Watch, HeartBeam).

SUMMARY:
The goal of this observational pilot study is to evaluate the investigational AK+ Guard™ software as a medical device (SaMD) for detection of moderate to severe hyperkalemia (serum potassium (K+) ≥ 6.5 mmol/L) in adults with chronic kidney disease (CKD).

Study objectives are:

* Arm 2A (Outpatient Diagnostic Accuracy): To generate a preliminary, real-world signal of the diagnostic performance of AK+ Guard™ when used in an ambulatory CKD cohort for identifying clinically significant hyperkalemia episodes (serum K+ ≥ 6.5 mmol/L) at the time of an outpatient laboratory draw.
* Arm 2B (Remote Patient Monitoring): To assess participant compliance, usability, and end-to-end system reliability of AK+ Guard™ when deployed for daily remote monitoring of CKD patients outside the clinical environment for up to four weeks.

DETAILED DESCRIPTION:
The AK+ Guard™ application is an investigational Software as a Medical Device (SaMD) developed by AccurKardia, Inc. (New York, USA). It is designed to aid in the diagnosis of moderate to severe hyperkalemia (serum potassium ≥ 6.5 mmol/L) in adults using artificial intelligence analysis of Lead I electrocardiogram (ECG) data. The software is intended as a clinical decision support tool for adults at risk of hyperkalemia, including but not limited to those with end-stage renal disease (ESRD), chronic kidney disease (CKD) on renin-angiotensin-aldosterone system inhibitors, heart failure, adrenal disorders, and patients taking aldosterone synthase inhibitors. The AK+ Guard™ application analyzes only Lead I ECG signals, which may be obtained from standard 12-lead ECGs, clinical-grade ECG devices with Lead I capability, or consumer wearable devices (e.g., Apple Watch).

This pilot study is designed to generate preliminary real-world evidence on both the diagnostic performance of the application and its usability in daily life. The study includes two arms:

Arm 2A - Outpatient Diagnostic Accuracy:

* Estimate sensitivity, specificity, PPV, and NPV of AK+ Guard™ in ambulatory CKD stages III-IV
* Evaluate interoperability across selected Lead I ECG capture devices (Apple Watch, HeartBeam, and 12 lead reference)
* Characterize system reliability metrics (upload success, algorithm runtime) in the outpatient setting

Arm 2B - Remote Patient Monitoring

* Quantify participant compliance, data completeness, and attrition during four week remote monitoring
* Evaluate user experience using System Usability Scale (SUS) score, Net Promoter Score (NPS), and semi structured feedback
* Capture technical performance metrics in a real world, unsupervised context

ELIGIBILITY:
Inclusion Criteria:

(Arm 2A - Outpatient Diagnostic Accuracy)

* Age 22 years or older
* CKD stages III-IV managed at Central Jersey Kidney Care outpatient clinic
* Scheduled outpatient serum potassium laboratory test
* On RAASi therapy or documented hyperkalemia (K+ ≥ 5.5 mmol/L) within the past 12 months
* Able to provide written informed consent

(Arm 2B - Remote Patient Monitoring)

* Completion of Arm 2A visit
* Owns an iPhone compatible with the study application

Exclusion Criteria (Both arms):

* Age 21 years or younger
* Pacemaker or implantable cardioverter defibrillator
* Pre existing Left Bundle Branch Block (LBBB), Right Bundle Branch Block (RBBB), Intraventricular Conduction Delay (IVCD), or clinically significant hypocalcemia
* Potassium lowering treatment administered before Lead I ECG acquisition
* Trauma, acute events, or active interventions altering potassium homeostasis
* Physical limitation precluding ECG acquisition

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adults aged 22 years or older with chronic kidney disease (CKD) stages III-IV who receive care at Central Jersey Kidney Care, an outpatient nephrology clinic. Eligible participants for Arm 2A will be identified at the time of a routine outpatient potassium blood draw. A subset of participants who complete Arm 2A will be invited to enroll in Arm 2B, which involves daily remote monitoring at home for up to four weeks. Participants must have an iPhone compatible with the study application to join Arm 2B.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Arm 2A: Sensitivity and specificity of AK+ Guard™ for detecting serum potassium greater than or equal to 6.5 mmol/L | Baseline (Day 0)
  Defined as serum K+ ≥ 6.5 mmol/L
Arm 2B: (a) Daily compliance rate (proportion of completed ECGs out of scheduled ECGs) | Daily monitoring up to 4 weeks (Day 28)
Arm 2B: (b) Mean System Usability Scale (SUS) score | Study completion at Week 4 (Day 28)
  10-item scale with final score between 0 and 100. The SUS score is an index of perceived usability (not a percentage), with higher scores indicating better usability. A score above 68 is generally considered above average usability, while lower scores suggest more usability concerns. The reported outcome will be the mean SUS score across participants.
Arm 2B: (c) Net Promoter Score (NPS) | Study completion at Week 4 (Day 28)
  Participant-reported likelihood of recommending the system to others, measured on a 0-10 scale, with higher scores indicating greater likelihood to recommend. Individual responses are converted into a Net Promoter Score (NPS), which ranges from -100 to +100. Positive values (>0) indicate overall customer loyalty and advocacy.

SECONDARY OUTCOMES:
Arm 2A: Positive Predictive Value (PPV) | Baseline (Day 0)
  Percentage (%) of positive hyperkalemia alerts generated by AK+ Guard™ that are confirmed as true positives by outpatient laboratory results.
Arm 2A: Negative Predictive Value (NPV) | Baseline (Day 0)
  Percentage (%) of negative results generated by AK+ Guard™ that are confirmed as true negatives by outpatient laboratory results.
Arm 2A: Device specific concordance | Baseline (Day 0)
  Percentage (%) of device-detected results that agree with outpatient laboratory results.
Arm 2A: Algorithm runtime | Baseline (Day 0)
  Time in seconds (s) required for the AK+ Guard™ algorithm to complete analysis, defined as the total of transmission time, processing time, and time to return results.
Arm 2A: Upload success rate | Baseline (Day 0)
  Percentage (%) of attempted ECG uploads that successfully complete without failure.
Arm 2B: Data completeness | Daily monitoring up to 4 weeks (Day 28)
  Percentage (%) of scheduled ECGs that are successfully completed.
Arm 2B: System reliability (application ("app") crash rate, upload failure less than 2 percent (%)) | Daily monitoring up to 4 weeks (Day 28)
Arm 2B: Number of service calls per participant | Daily monitoring up to 4 weeks (Day 28)
Arm 2B: False positive alarm rate (less than 20%) | Daily monitoring up to 4 weeks (Day 28)
  Percentage (%) of alarms generated by AK+ Guard™ that are not confirmed as true clinical events by outpatient laboratory results.

OTHER OUTCOMES:
Arm 2A (Exploratory): Sensitivity (stratified) | Baseline (Day 0)
  Sensitivity of AK+ Guard™ for detecting serum K+ ≥ 6.5 mmol/L, stratified by CKD stage, renin-angiotensin-aldosterone system inhibitor (RAASi) use, and comorbidity profile. Reported as point estimate (%) with confidence interval.
Arm 2A (Exploratory): Positive Predictive Value (PPV, stratified) | Baseline (Day 0)
  PPV of AK+ Guard™ for detecting serum K+ ≥ 6.5 mmol/L, stratified by CKD stage, renin-angiotensin-aldosterone system inhibitor (RAASi) use, and comorbidity profile. Reported as point estimate (%) with confidence interval.
Arm 2A (Exploratory): Negative Predictive Value (NPV, stratified) | Baseline (Day 0)
  NPV of AK+ Guard™ for detecting serum K+ ≥ 6.5 mmol/L, stratified by CKD stage, renin-angiotensin-aldosterone system inhibitor (RAASi) use, and comorbidity profile. Reported as point estimate (%) with confidence interval.
Arm 2B (Exploratory): Participant perception of medication safety | Baseline (Day 0) and at study completion (Day 28)
  Change from baseline in survey responses on perceived benefit of AK+ Guard™ for monitoring potassium and identifying dangerous levels earlier. Each item is rated on a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree).
Arm 2B (Exploratory): Participant anxiety and comfort | Baseline (Day 0) and at study completion (Day 28)
  Change from baseline in survey responses on reassurance and anxiety, and comfort with using AK+ Guard™. Each item is rated on a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Central Jersey Kidney Care - Hypertension & Nephrology Associates, Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided